Study title: Aspirin Prescription For Moderate- and High-Risk Obstetric Population in Outpatient Clnic; A Quality Improvement Project.

Date: 4/11/2024

NCT06694233

# **CLINICAL AUDIT PROJECT PLAN**

Please complete this project plan before starting your project.

1. Short Title of Audit: Aspirin Prescription For Moderate- and High-Risk Obstetric Population

in Outpatient Clnic; A Quality Improvement Project.

### 2. Details of Audit Lead

| Audit Lead: | Name: Islam Elkhateb | Designation: Registrar |
|---|---|---|
| Contact details: | E-mail: islamtarekhamed@gmail.com | Phone: 99780408 |

#### 3. Details of Audit Sponsor:

| | Name: | Designation: Consultant |
|----------------|-------|---------------------------------|
| Audit Sponsor: | Name: | Designation: Consultant |
| | Name: | Designation: Head of department |

4. Date plan completed: 27/10/2024

### 5. Rationale and Objectives of the Audit:

Preeclampsia is a syndrome characterized by the new onset of hypertension plus proteinuria, end-organ dysfunction, or both after 20 weeks of gestation. It complicates 3-5% of pregnancies.

Low-dose aspirin reduces the frequency of preeclampsia, as well as related adverse pregnancy outcomes (preterm birth, growth restriction), by 10 to 70 percent when taken by patients at moderate to high risk of the disease. It has an excellent maternal/fetal safety profile, thus it is a reasonable preventive strategy for these patients.

A pilot study at our hospital found that not all patients who are candidates for aspirin prescription receive it. The aim of this audit cycle is to increase aspirin prescription rates for moderate and high risk obstetric population.

### 6. Based on your audit rationale how would you classify this audit?

| This is an external audit ☐ (e.g. National audit) | This is an internal audit √ (e.g arising from Trust objectives/ risks/ incidents / complaints/ NICE guidelines compliance etc) |
|---|---|
| This a Division/Service priority | This is an individual clinician interest $\Box$ |
| (e.g. part of Divisional or Team Service improvement priorities) | (e.g. personal interest, personal development or as part of an educational or training programme) |

#### 7. What criteria will be audited?

| Criterion (suggested proforma) | Current | Target | Exception | Evidence |
|--------------------------------|---------|--------|-----------|----------|
| Constitution (Constitution) | | 3.0 | | |

| Advise pregnant women at high risk of pre-eclampsia to take 75 mg to 150 mg of aspirin daily from 12 weeks until the birth of the baby. Women at high risk are those with any of the following: 1. hypertensive disease during a previous pregnancy 2. chronic kidney disease 3. autoimmune disease such as systemic lupus erythematosus or antiphospholipid syndrome 4. type 1 or type 2 diabetes 5. chronic hypertension. [2010, amended 2019] Advise pregnant women with more than 1 moderate risk factor for pre-eclampsia to take 75 mg to 150 mg of aspirin daily from 12 weeks until the birth of the baby. Factors indicating moderate risk are: 1. nulliparity 2. age 40 years or older 3. pregnancy interval of more than 10 years 4. body mass index (BMI) of 35 kg/m2 or more at first visit 5. family history of pre-eclampsia 6. multi-fetal pregnancy. [2010, amended 2019] | 40% | 100% | None | Hypertension<br>in pregnancy:<br>diagnosis and<br>management.<br>NICE guideline<br>133. Last<br>updated 17<br>April 2023. |
|---|---|---|---|---|
|---|---|---|---|---|

# 8. How will you implement changes and recommendations?

- Labels/ reminders maybe put posted in outpatient department rooms/ clinics.
- Proforma/ labels maybe put in each patient file (like the VTE risk assessment table)
- The topic will be mentioned in the morning meeting.
- The topic maybe covered and illustrated in one of the biweekly scientific meetings.
- An email message maybe sent to all teams on the OBGYN department group.

# 9. Do the audit standards cover the practice of one or more professional groups?

| This is a Multi-disciplinary audit | This is an Uni-disciplinary audit | √ |
|------------------------------------|-----------------------------------|---|
|------------------------------------|-----------------------------------|---|

# 10. What data collection method will be used?

Concurrent and prospective data collection: Aspirin presciprion rates for high- and moderate- risk groups over the month of October were investigated.

After drawing receommendations and implementing changes, Aspirin prescription rates over the next six months (November 2024- April 2025) will be monitored and audited.

# 11. What is your sample size?

Interval sampling is the method used for sample size calculation in this audit, in which all cases who will present in May 2025 will be included.

# 12. What is your planned project timetable

| Project Activity | Estimated Completion Date |
|---|---|
| Date of completiomn of data collection, inputting, and analysis | 31/10/2024 |
| Proposed date for presentation of results and recommendations for the modification of practice | 4/11/2024 |
| Proposed date for start of implementation of modifications | 5/11/2024 |
| Proposed date for re-auditing the results | 5/ 2025 |

| 40 | 11 | | | | L a : | : اممیرام | 41- :- | |
|---|---|---|---|---|---|---|---|---|
| 13 | . HOW W | ill service | users o | or carers | pe inv | oivea i | n this | audit ? |

| Service users are not be involved in this audit since they cannot modify/ control the outcome. |
|---|

| Project lead: | Project supervisors: |
|------------------|----------------------|
| Department head: | |